CLINICAL TRIAL: NCT02833415
Title: Visceral Adiposity and Diabetes: Translating Form to Function Using Imaging
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Ian Neeland, M.D., University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: STU-012015-064; K23DK106520 (NIH)
Record Dates: First submitted 2016-07-05; First posted 2016-07-14 (Estimated); Results first posted 2019-05-02 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Obesity, Visceral
Keywords: Visceral; Obesity; Adipose; Diabetes
MeSH Terms: conditions — Obesity, Abdominal; Obesity; Diabetes Mellitus | interventions — Glycerol; empagliflozin; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Empagliflozin (Experimental): Empagliflozin 10 mg by mouth daily for 3 months.
  Interventions: Drug: [U-13C3] glycerol; Drug: Empagliflozin
- Placebo (Placebo Comparator): Placebo one tablet daily for 3 months
  Interventions: Drug: [U-13C3] glycerol; Drug: Placebo (for Empagliflozin)

INTERVENTIONS:
Drug: [U-13C3] glycerol — Ingestion of [U-13C3] glycerol based on human's body weight such as (50 mg/kg body weight).
  Other Names: Glycerine; Glycerin
Drug: Empagliflozin — Active drug
  Other Names: EMPA; Jardiace
  Arms: Empagliflozin
Drug: Placebo (for Empagliflozin) — Placebo tablet manufactured to mimic EMPA 10 mg tablet.
  Other Names: Placebo; Sugar pill
  Arms: Placebo

SUMMARY:
This study is a clinical study to investigate the gluconeogenesis pathway related to visceral adipose tissue (VAT) in obese individuals without type 2 diabetes and the effects of empagliflozin (EMPA) on glucose homeostasis in viscerally-obese individuals using functional studies of glycerol metabolism in hepatic gluconeogenesis using a well-validated nuclear magnetic resonance (NMR) spectroscopy platform.

DETAILED DESCRIPTION:
Diabetes mellitus type II is the consequence of insulin resistance and pancreatic beta cell failure resulting from a variety of metabolic insults, one of which is excess body adiposity/obesity. In the diabetic individual, hepatic gluconeogenesis may go uninhibited due to failure of the body's normal feedback mechanisms to appropriately incorporate glucose into cells via insulin signaling, leading to excess gluconeogenesis and hyperglycemia. The substrate for this excess glucose derives from multiple sources in the liver including dietary glycerol, adipose-derived glycerol from lipolysis, and substrates from the citric acid cycle. In the normal state, lipolysis is maintained at a steady state in equilibrium between stored dietary triglycerides and free fatty acids. However, in situations of triglyceride excess (e.g. in the obese state), lipolysis may become overactive resulting in increased free fatty acids and adipose-derived glycerol. This excess glycerol drives hepatic gluconeogenesis and is incorporated into glucose and released into the blood, leading to hyperglycemia, and ultimately diabetes and its clinical sequelae.

A popular hypothesis linking visceral fat with excess gluconeogenesis is delivery of glycerol arising from mesenteric triglyceride turnover directly into the portal circulation and to the liver. Glycerol is a primary substrate for gluconeogenesis in the liver. Under normal conditions, hepatic gluconeogenesis begins from glycerol ingested in the diet which is converted to glycerol-3-phosphate and subsequently dihydroxyacetone phosphate (DHAP) in the liver. DHAP is converted to fructose-1,6-bisphosphate which undergoes a series of reactions to become a single 6-carbon glucose molecule. Adipocytes contribute glycerol to hepatic gluconeogenesis through lipolysis of triglyceride stores. Although glycerol-gluconeogenesis has been extensively studied in animals, the traditional reliance on radioactive tracers makes translation to humans difficult for many reasons. We aim to use new techniques to explore the mechanisms behind altered glucose metabolism related to excess visceral adiposity in obese adults by quantifying the relative contributions of varying substrates to liver-derived glucose. One such method uses 13C3 labeled glycerol to trace the incorporation of glycerol from dietary sources to hepatic gluconeogenesis. This technology utilizes nuclear magnetic resonance (NMR) spectroscopy, a technique that does not require ionizing radiation and has been extensively validated, to analyze the NMR spectra of plasma glucose and quantify the "percent enrichment" of the circulating glucose molecules with labeled glycerol. In turn, differences in enrichment reflect variability in hepatic glucose metabolism as it relates to the contribution of glycerol from visceral adipose tissue to gluconeogenesis.

The rationale of this project is to utilize existing technology to investigate the impact of excess visceral adiposity on glycerol metabolism in hepatic gluconeogenesis in obese adults without diabetes and to explore the effects of treatment with EMPA on visceral adiposity related glucose homeostasis.

ELIGIBILITY:
Inclusion Criteria:

* Obese, defined as BMI ≥ 30 kg/m2, at both time of abdominal fat imaging and at study entry.
* Ages 30-65
* No prevalent diagnosis of type 2 diabetes mellitus, either at the time of abdominal fat imaging or at study entry.
* Previous abdominal fat quantification by magnetic resonance imaging in the Dallas Heart Study or possible neck-to-knee MRI for VAT measurement may be performed.

Exclusion Criteria:

* Pregnant or breastfeeding
* Incarcerated
* Chronic kidney or liver disease
* History of frequent (>2/year) urinary tract infections
* Non-obese either at time of abdominal fat imaging or at present.
* Greater than 10% change in body weight (kg) between time of abdominal fat imaging and present.
* Has donated blood within last 6 weeks
* Cannot give informed consent, understand the protocol, or tolerate any aspect of the protocol
* If undergoing MRI, persons with metal implants contraindicated for 3Tesla MRI exams will be excluded. Severe claustrophobia will also be assessed prior to an MRI exam.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-03; Primary Completion 2018-01 (Actual); Study Completion 2018-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ian Neeland, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD sharing will be done upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Access Criteria: Email the PI with request.

REFERENCES:
- [Background] Neeland IJ, Ayers CR, Rohatgi AK, Turer AT, Berry JD, Das SR, Vega GL, Khera A, McGuire DK, Grundy SM, de Lemos JA. Associations of visceral and abdominal subcutaneous adipose tissue with markers of cardiac and metabolic risk in obese adults. Obesity (Silver Spring). 2013 Sep;21(9):E439-47. doi: 10.1002/oby.20135. Epub 2013 May 19. PMID 23687099
- [Background] Neeland IJ, Turer AT, Ayers CR, Powell-Wiley TM, Vega GL, Farzaneh-Far R, Grundy SM, Khera A, McGuire DK, de Lemos JA. Dysfunctional adiposity and the risk of prediabetes and type 2 diabetes in obese adults. JAMA. 2012 Sep 19;308(11):1150-9. doi: 10.1001/2012.jama.11132. PMID 22990274
- [Background] Nurjhan N, Kennedy F, Consoli A, Martin C, Miles J, Gerich J. Quantification of the glycolytic origin of plasma glycerol: implications for the use of the rate of appearance of plasma glycerol as an index of lipolysis in vivo. Metabolism. 1988 Apr;37(4):386-9. doi: 10.1016/0026-0495(88)90140-0. PMID 3357420
- [Background] Baba H, Zhang XJ, Wolfe RR. Glycerol gluconeogenesis in fasting humans. Nutrition. 1995 Mar-Apr;11(2):149-53. PMID 7647479
- [Background] Jin ES, Sherry AD, Malloy CR. Interaction between the pentose phosphate pathway and gluconeogenesis from glycerol in the liver. J Biol Chem. 2014 Nov 21;289(47):32593-603. doi: 10.1074/jbc.M114.577692. Epub 2014 Oct 6. PMID 25288790
- [Derived] Neeland IJ, de Albuquerque Rocha N, Hughes C, Ayers CR, Malloy CR, Jin ES. Effects of Empagliflozin Treatment on Glycerol-Derived Hepatic Gluconeogenesis in Adults with Obesity: A Randomized Clinical Trial. Obesity (Silver Spring). 2020 Jul;28(7):1254-1262. doi: 10.1002/oby.22854. PMID 32568464

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Empagliflozin | Placebo
Started | 20 | 20
Completed | 18 | 17
Not Completed | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Empagliflozin | Placebo | Total
Number analyzed (Participants) | 18 | 17 | 35
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 50.5 [43 to 56] | 54 [48 to 59] | 53 [46 to 59]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 22
  Male | 7 | 6 | 13
Race/Ethnicity, Customized [Number; unit: participants]
  African-American | 5 | 7 | 12
Systolic Blood Pressure [Median (Inter-Quartile Range); unit: mmHg] | 126 [117 to 138] | 132 [127 to 141] | 130 [120 to 139]
Hemoglobin A1C [Median (Inter-Quartile Range); unit: percent of glycosylated hemoglobin] | 5.6 [5.4 to 5.9] | 5.9 [5.6 to 6.1] | 5.8 [5.4 to 6.0]
Body Mass Index [Median (Inter-Quartile Range); unit: kg/m^2] | 36.8 [32.9 to 38.8] | 35.3 [32.7 to 39.6] | 35.5 [32.9 to 39.6]
Visceral Fat [Median (Inter-Quartile Range); unit: kg] | 5.4 [4.0 to 7.3] | 4.3 [3.8 to 6.7] | 5.4 [3.9 to 7.2]

OUTCOME MEASURES:

1. Primary Outcome: Change in Glycerol Enrichment
Description: [U-13C3] glycerol enrichment in plasma blood glucose over time will be measured by nuclear magnetic resonance spectroscopy. This is a percentage change from baseline to follow up in the percent enrichment of exogenous glycerol in blood glucose. We are unable to report a measure of central tendency and dispersion as the outcome is a percent change in the area under the enrichment curve for each group between baseline and follow-up. There is no measure of central tendency for these measurements without bootstrapping, which was not performed.
Time Frame: 3 months
Measure: Number; unit: Percentage change
Arm/Group | Empagliflozin | Placebo
Number analyzed (Participants) | 18 | 17
Percentage change | 6.5 | 1.4
Statistical Analysis 1: Comparison: Empagliflozin; Baseline to Followup; Test type: Other — Differences of Least Squares Means; p = 0.0053, Mixed Models Analysis; Differences of Least Squares Means = 0.9398, Standard Error of Mean 0.2941
Statistical Analysis 2: Comparison: Placebo; Baseline to Followup; Test type: Other — Differences of Least Squares Means; p = 0.5394, Mixed Models Analysis; Differences of Least Squares Means = 0.1520, Standard Error of Mean 0.2424

ADVERSE EVENTS:
Time Frame: 3 months
Description: Adverse Events Definition: Any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research.
Groups:
- Empagliflozin: Empagliflozin 10 mg daily by mouth
- Placebo: Placebo daily by mouth
Arm/Group | Empagliflozin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 1/20 | 0/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Empagliflozin (N=20) | Placebo (N=20)
Urinary Tract Infection (Renal and urinary disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-13): https://cdn.clinicaltrials.gov/large-docs/15/NCT02833415/Prot_SAP_000.pdf